CLINICAL TRIAL: NCT01851421
Title: Fat Metabolism and Function Altering Polymorphisms in MC3R
Brief Title: Fat Metabolism and Melanocortin 3 Receptors in African Americans
Status: Terminated | Type: Observational
Why Stopped: Slow/Insufficient accrual
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130097; 13-CH-0097
Record Dates: First submitted 2013-05-09; First posted 2013-05-10 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Obesity; Healthy Volunteers
Keywords: Lipogenesis; Adult; Obesity; LIPOLYSIS; Melanocortin-3 Receptor
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, genomic DNA (extracted from whole blood)

GROUPS / COHORTS (2):
- Double-Variant MC3R: Volunteers with homozygous polymorphisms causing protein changes to T6K and V81I.
- Wild Type MC3R: Volunteers with no polymorphisms in MC3R gene.

SUMMARY:
Background:

- Melanocortin receptors are proteins in the body that help send messages between body systems. One such receptor, the melanocortin 3 receptor (MC3R), is important for regulating body weight. Differences in MC3R can affect fat metabolism - or how the body handles fat. Some people who have changes in the MC3R genetic code are heavier than those who do not have these changes. These changes are found more often in African Americans. Researchers want to study the MC3R in African American adults to see how these changes may affect fat metabolism. They will look at overweight adults with either the most common genetic code for the MC3R or a rare variant.

Objectives:

- To study the role of the MC3R in body weight and fat metabolism.

Eligibility:

* Healthy African American volunteers between 18 and 55 years of age.
* Volunteers must be overweight (body mass index at least 30 kg/m2) but weigh less than 450 lbs.

Design:

* The study consists of an outpatient screening visit and a 7-day inpatient visit with dietary studies.
* Participants will be screened with a physical exam and medical history. Blood samples will be collected. (Participants will need to fast for 10 hours before giving blood samples.) A body scan will be given to determine fat, bone, and muscle content. Participants will complete a 3-day dietary assessment to record their food and drink consumption. They will also have an exercise test to look at heart and lung function.
* Participants will have a 7-day inpatient stay. They will have a regular diet for the first 3 days of the study. For the final 4 days, they will have a diet with a higher fat content.
* During the inpatient visit, participants will have the following study procedures:
* Body measurements
* Daily exercise routine
* Imaging studies of the body
* Measurement of a whole day s energy expenditure (spending one day in metabolic chamber-day 5)
* Frequent blood samples
* Urine collection for 24 hours (days 3 and 7)
* Fat biopsy (collection of a small sample of fat tissue from under the skin on the abdomen)
* Insulin and metabolism tests while eating the two different diets (day 4 and day 7).
* After the final insulin and metabolism test, participants will be discharged from the study.

DETAILED DESCRIPTION:
Our prior studies have found that children with homozygosity for two rare Melanocortin 3 Receptor (MC3R) polymorphisms (T6K+V81I) have greater fat mass compared to wild type children. These polymorphisms are about 10-fold more prevalent in Non-Hispanic Black than White Americans. In vitro, T6K+V81I causes MC3R hypofunction. Since mouse models and limited human data suggest the MC3R may be involved in regulating substrate oxidation, and therefore fatty acid disposal, we propose to study 30 Non-Hispanic Black BMI-matched subjects with homozygous T6K+V81I or wild-type MC3R to compare substrate turnover (fatty acids and glucose) during fasting and under conditions of hyperinsulinemia after adaptation from a normal-fat to a high-fat isocaloric diet. Using adipocytes obtained from biopsies, we will also study glucose and fatty acid uptake, storage and mobilization in vitro. We hypothesize that this study will shed light on the role of the MC3R in substrate metabolism and energy expenditure, and will yield information that may assist in the development of more effective approaches for the treatment of obesity in Non-Hispanic Black Americans.

ELIGIBILITY:
* INCLUSION CRITERIA

Volunteers will qualify if they meet the following criteria

1. Age 18-55 years. Subject age is limited to 55y maximum because subjects are required to complete a maximal exercise test as part of their evaluations. Studying only younger patients decreases the risks of such exercise tests.
2. Non-Hispanic Black by self-identification with (to the best of the subject s knowledge) all 4 grandparents considered Non-Hispanic Black. Because T6K+V81I MC3R is 10-times more prevalent among Non-Hispanic Blacks, only Non-Hispanic Blacks will be eligible to participate.
3. Obesity, defined as body mass index (BMI) greater than or equal to 30 kg/m2 and weight under 450 lbs, in order for subjects to be able to undergo DXA scanning.
4. Willing to undergo genetic screening to establish that subject is either homozygous wild type for MC3R or homozygous for T6K+V81I MC3R, with the absence of other genetic causes of monogenic obesity (for both study and control groups).
5. Good general health. In general, subjects should take no medications. However, individuals taking medications for obesity-related co-morbid conditions, who have not had changes in dosage for more than 6 months, may be included, at the discretion of the principal investigator.
6. For females, a negative pregnancy test at the initial evaluation. Because pregnancy is a state in which weight gain is expected and appropriate, pregnant individuals would not be suitable for this study. Sexually active women must be using an effective form of birth control. These methods include abstinence, oral contraceptives, an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended (One of these methods must have been used by the subject for at least two months prior to the start of the study).

EXCLUSION CRITERIA

Volunteers will be excluded (and referred to non-experimental treatment programs as needed) for the following reasons:

1. Subjects with a major medical illnesses that in the opinion of the medical team would impede interpretation of results, including significant renal, hepatic (other than obesity-related steatosis), gastrointestinal, most endocrinologic (e.g., Cushing syndrome, untreated hyper- or hypothyroidism, pheochromocytoma), hematological problems (e.g. -PT/PTT values that are prolonged greater than or equal to 3 seconds from the upper limit of the normal or thrombocytopenia < 70,000) or pulmonary disorders; or porphyria;
2. Current users of tobacco products;
3. Subjects following a diet with specific food requirements such as vegetarian, vegan, or kosher;
4. Women who are pregnant or who are currently nursing an infant or have irregular menses;
5. Individuals who have current substance abuse or a psychiatric disorder or other condition that in the opinion of the investigators would impede competence or adherence;
6. Recent (3 months) use of anorexiant medications;
7. Subjects using medications known to affect glucose and fatty acid metabolism and/or absorption;
8. Subjects on anticoagulatns, or those who cannot safely stop NSAIDs or antiplataelet agents for 10 days (a week prior to and three days after their biopsy)
9. Subjects with weight change of more than 3% of body weight in the past two months;
10. Subjects currently using a weight loss diet;
11. Subjects with untreated hypertension: a consistently (2 weeks apart) elevated systolic blood pressure of greater than 160 mm Hg and/or a diastolic flood pressure greater than 95 mm Hg.
12. Subjects with a history of keloid formation, since such individuals may have greater scarring after biopsies or intravenous catheter placement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Comunity sample
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Free fatty acid reflux rate measured on a high- fat diet during the hyperinsulinemic state | 3 hours
  FFA flux by isotopic study

SECONDARY OUTCOMES:
Free fatty acid flux rate in the post-absorptive state and estimates of whole body glucose disposal and endogenous glucose production assessed during postabsorptive and hyperinsulinemic states on both diets | 4 days
  FFA flux by isotopic study

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Feng N, Young SF, Aguilera G, Puricelli E, Adler-Wailes DC, Sebring NG, Yanovski JA. Co-occurrence of two partially inactivating polymorphisms of MC3R is associated with pediatric-onset obesity. Diabetes. 2005 Sep;54(9):2663-7. doi: 10.2337/diabetes.54.9.2663. PMID 16123355
- [Background] Lee B, Koo J, Yun Jun J, Gavrilova O, Lee Y, Seo AY, Taylor-Douglas DC, Adler-Wailes DC, Chen F, Gardner R, Koutzoumis D, Sherafat Kazemzadeh R, Roberson RB, Yanovski JA. A mouse model for a partially inactive obesity-associated human MC3R variant. Nat Commun. 2016 Jan 28;7:10522. doi: 10.1038/ncomms10522. PMID 26818770
- [Background] Demidowich AP, Parikh VJ, Dedhia N, Branham RE, Madi SA, Marwitz SE, Roberson RB, Uhlman AJ, Levi NJ, Mi SJ, Jun JY, Broadney MM, Brady SM, Yanovski JA. Associations of the melanocortin 3 receptor C17A + G241A haplotype with body composition and inflammation in African-American adults. Ann Hum Genet. 2019 Sep;83(5):355-360. doi: 10.1111/ahg.12315. Epub 2019 Apr 2. PMID 30937899
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-CH-0097.html